CLINICAL TRIAL: NCT00006456
Title: Fractionated Stereotactic Body Radiosurgery for Extracranial Tumors
Brief Title: Stereotactic Radiosurgery in Treating Patients With Liver Metastases, Lung Metastases, or Other Advanced Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Danny Song, MD, Virginia Commonwealth University/Massey Cancer Center
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068151; P30CA016059 (NIH); MCV-MCC-9812-2C; NCI-V00-1612
Record Dates: First submitted 2000-11-06; First posted 2003-01-27 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; lung metastases; liver metastases
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: stereotactic radiosurgery

SUMMARY:
RATIONALE: Stereotactic radiosurgery delivers x-rays directly to the tumor and may cause less damage to normal tissue.

PURPOSE: Phase II trial to study the effectiveness of stereotactic radiosurgery in treating patients who have liver metastases, lung metastases, or other advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of fractionated stereotactic body radiosurgery in patients with advanced extracranial tumors.
* Assess the toxicities of this treatment regimen in these patients.
* Determine tumor response and cause of death in these patients treated with this regimen.

OUTLINE: Patients receive fractionated stereotactic body radiosurgery over 30 minutes for 5-10 days for a total of 3 treatments.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 10-25 patients will be accrued within 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignancy

  * Extracranial recurrent or metastatic disease or primary tumor not predicted to be controlled with standard radiotherapy
  * Incurable with any standard therapy
* No tumors involving critical structures (e.g., mucosal surfaces (bowel or bladder) or heart)
* Tumor visible by CT scan

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 2.0 times upper limit of normal (ULN)
* AST and ALT less than 5 times ULN

Renal:

* Creatinine less than 2.0 mg/dL

Pulmonary:

* FEV1 greater than 0.75 L

Other:

* No unsuitable size or geometric proportion that would preclude stereotactic immobilization
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 14 days since prior anticancer biologic therapy and recovered

Chemotherapy:

* At least 14 days since prior anticancer chemotherapy and recovered

Endocrine therapy:

* At least 14 days since prior anticancer endocrine therapy and recovered

Radiotherapy:

* See Disease Characteristics
* At least 14 days since prior anticancer radiotherapy and recovered

Surgery:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 1999-02; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danny Y. Song, MD, Study Chair — Massey Cancer Center
Locations (1):
- Massey Cancer Center, Richmond, Virginia, United States